CLINICAL TRIAL: NCT07188701
Title: The Effect of an Exercise Program Applied Through Telerehabilitation on Pain, Sleep Quality, Depression, Anxiety, and Stress in Individuals With Chronic Non-specific Neck Pain
Brief Title: Telerehabilitation Exercise Program for Individuals With Chronic Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGU-FTR-DT-01; IGU-FTR-DT-01 (Other: Istanbul Gelisim University)
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Non-Specific Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Telerehabilitation Exercise Program (Experimental): Participants received a 6-week structured telerehabilitation exercise program delivered via Zoom under the supervision of a physiotherapist. The program was performed 4 days per week, approximately 20-30 minutes per session, focusing on posture correction, cervical stabilization, mobility, and pain management strategies
  Interventions: Behavioral: Telerehabilitation Exercise Program
- Active Comparator: Home Exercise Program (Active Comparator): Participants received a 6-week home exercise program. Exercises were demonstrated once weekly via Zoom by a physiotherapist. Participants performed the program independently at home, 4 days per week, 20-30 minutes per session.
  Interventions: Behavioral: Telerehabilitation Exercise Program

INTERVENTIONS:
Behavioral: Telerehabilitation Exercise Program — 1. Telerehabilitation Exercise Program
     Intervention Description:
     "A 6-week structured telerehabilitation exercise program delivered via Zoom under the supervision of a physiotherapist. Sessions were conducted 4 days per week, approximately 20-30 minutes each. Exercises focused on posture correction, cervical stabilization, mobility, and pain management strategies."
  2. Home Exercise Program
  Intervention Description:
  "A 6-week home exercise program for chronic non-specific neck pain. Exercises were demonstrated once weekly via Zoom by a physiotherapist, and participants performed them independently at home on the remaining days. Each session lasted 20-30 minutes and included stretching, strengthening, and posture training."
  Other Names: Online Physiotherapy

SUMMARY:
This study examined whether a 6-week telerehabilitation exercise program could reduce pain and improve daily functioning in people with chronic non-specific neck pain. Participants were adults aged 18-65 who had neck pain for at least 3 months. The program included guided physiotherapy-based exercises delivered online using video calls. Outcomes measured included pain intensity, disability, mood, and sleep quality. The goal was to evaluate if telerehabilitation is an effective and safe method for managing chronic neck pain.

DETAILED DESCRIPTION:
Chronic non-specific neck pain is a common condition that negatively affects quality of life and daily functioning. Conventional rehabilitation programs often require face-to-face sessions, which may be limited by access barriers. Telerehabilitation offers a practical alternative by providing physiotherapy interventions remotely through online platforms.

This study investigated the effects of a 6-week telerehabilitation-based exercise program on individuals with chronic non-specific neck pain. Participants were randomly assigned to groups and received structured exercise sessions guided by a physiotherapist via video calls. Primary outcome was pain intensity measured with the Visual Analog Scale (VAS). Secondary outcomes included disability assessed by the Neck Disability Index (NDI), mood and psychological well-being assessed with the Beck Depression Inventory (BDI-21) and Depression Anxiety Stress Scale (DASS-21), and sleep quality measured with the Pittsburgh Sleep Quality Index (PSQI).

The objective was to evaluate whether telerehabilitation exercises can reduce pain and disability, and improve psychological health and sleep quality, providing evidence for its effectiveness as a non-invasive and accessible management strategy for neck pain.

ELIGIBILITY:
Inclusion Criteria:Aged 18-55 years

History of neck pain lasting at least 3 months

Willingness to participate in the study

Having an active internet connection and access to a tablet or computer at home

Ability to read and write in Turkish

-

Exclusion Criteria:

* Traumatic cervical injuries

Tumoral conditions

Cognitive impairments

Receiving physiotherapy for neck pain within the last 6 months

Presence of visual or hearing impairments

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | Baseline and after 6 weeks of intervention
  Change in pain intensity assessed by the Visual Analog Scale (VAS). Scores range from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Neck Disability (NDI) | Baseline and after 6 weeks of intervention
  Change in functional disability assessed by the Neck Disability Index (NDI). Scores range from 0 to 50, with higher scores indicating greater disability.
Sleep Quality (PSQI) | Baseline and after 6 weeks of intervention
  Change in sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI). Scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Depression, Anxiety, and Stress (DASS-21) | Baseline and after 6 weeks of intervention
  Change in psychological outcomes assessed by the Depression, Anxiety, Stress Scale (DASS-21). Subscale scores range from 0 to 42.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Gelişim University, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valenza-Pena G, Calvache-Mateo A, Valenza MC, Granados-Santiago M, Raya-Benitez J, Cabrera-Martos I, Diaz-Mohedo E. Effects of Telerehabilitation on Pain and Disability in Patients with Chronic Neck Pain: A Systematic Review and Meta-Analysis. Healthcare (Basel). 2024 Apr 6;12(7):796. doi: 10.3390/healthcare12070796. PMID 38610217
- See also: Official website of Istanbul Gelişim University, the institution where the study is conducted. — https://gelisim.edu.tr/